CLINICAL TRIAL: NCT04421651
Title: Dance Movement Therapy in the Treatment of Depressed Patients: A Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jyvaskyla (Other)
Collaborators: The Social Insurance Institution of Finland (Unknown); Finnish Dance Therapy Association (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UJyvaskyla DMT trial
Record Dates: First submitted 2020-05-25; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Depression
Keywords: Dance Movement Therapy; Adults; Depression; Beck Depression Inventory; Clinical Outcomes in Routine Evaluation - Outcome Measure; The Symptoms Check List-90
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): The participants in the treatment group were offered 20 Dance movement therapy sessions in addition to standard care.
  Interventions: Behavioral: Dance Movement Therapy group
- Control group (No Intervention): Participants in the control group continued treatment as usual in the health services.

INTERVENTIONS:
Behavioral: Dance Movement Therapy group — DMT-intervention was facilitated by a dance movement therapist and included 20 x 75 mins sessions within 10 weeks.
  Arms: Treatment group

SUMMARY:
This multi-centre research investigates the effects of dance movement therapy (DMT) on participants diagnosed with depression. In total, 109 persons participated in the study in various locations in Finland. All participants received treatment as usual (TAU). They were randomised into DMT + TAU (n = 52) or TAU-only (n = 57). The participants in the DMT + TAU group were offered 20 DMT sessions twice a week for 10 weeks in addition to standard care. The measurement points included pre-treatment measurement at the baseline and post-treatment measurement at the end of the intervention, which was 10 weeks after the pre-treatment measurement. The follow-up measurement was 3 months after the post-treatment measurement. The effects of the intervention were assessed with a clinical measure of depression (BDI-I) and with indicators of physical and psychological distress (CORE-OM and SCL-90). The participants in the treatment group (DMT+TAU) were compared to the participants in the control group who received TAU-only.

DETAILED DESCRIPTION:
This research investigates the outcomes of dance movement therapy (DMT) groups in the treatment of adults with depression. In total, 157 participants were involved. Of them, 109 were randomized into DMT group (n = 52) or control group (n = 57). The rest of the participants participated in non-randomized DMT groups. All participants met the criteria for the eligibility for rehabilitation psychotherapy, had depression diagnosed by a doctor, and the severity of depression threatened the ability to work/ study. All participants received treatment as usual during the research. DMT-intervention was facilitated by a dance movement therapist and included 20 x 75 mins sessions within 10 weeks. Depressive symptoms (BDI), physical and psychological distress (CORE-OM, SCL-90), ability to work/study, and body image were assessed at three measurement points: pre-measurement at the baseline, post-measurement 10 weeks after the pre-treatment measurement, and a follow-up measurement three months after the post-treatment measurement.

This research includes a larger number of participants (N = 109) than have been involved in previous studies utilising randomised controlled trials in research designs. The research generates further information about the effectiveness of dance movement therapy groups in the rehabilitation of depression as it was conducted in five cities across Finland. This type of multi-centre research can provide a realistic picture of the typical practice of a range of dance movement therapists working with participants in various geographic locations.

ELIGIBILITY:
Inclusion Criteria:

* The participant needed to have a diagnoses of depression by a psychiatrist or general practitioner (ICD -diagnostic system). The researchers checked that the participants were working age (18-65 years of age) and fulfilled the criteria for rehabilitative psychotherapy in Finland: at least three months of relevant treatment since depression was diagnosed; the participants' ability to work or study is impaired by depression; a psychiatrist has determined that rehabilitative psychotherapy is necessary to improve or support the participant's ability to work or study.

Exclusion Criteria:

* active suicidal ideation; psychotic symptoms; substance misuse that is on a critical level. Also, interviewees who had pain-related problems that restricted daily life or were pregnant were not admitted to the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline depressive symptoms (Beck Depression Inventory; BDI) at 10-week post-treatment measurement | 10 weeks
  BDI measures depressive symptoms with 21 items. Each item is scored 0-3 and sum scores are calculated on the basis of participants' responses. The total sum score can range from 0 to 63.
Change from post-treatment depressive symptoms (Beck Depression Inventory; BDI) at three-month follow-up measurement | 3 months
  The change in depressive symptoms between the post-treatment measurement at the end of the 10-week intervention and the 3-month follow-up.

SECONDARY OUTCOMES:
Change from baseline psychological distress (Clinical Outcomes in Routine Evaluation - Outcome Measure; CORE-OM) at 10-week post-treatment measurement | 10 weeks
  The CORE-OM comprises 43 items and four dimensions of well-being, problems, life functioning, and risk for aggressive/suicidal behaviour. Each item is scored from 0 to 4. CORE-OM items are summed and then divided by the number of answered items, which is then multiplied by ten; that is, the total scores ranges from 0 to 40.
Change from post-treatment psychological distress (Clinical Outcomes in Routine Evaluation - Outcome Measure; CORE-OM) at three-month follow-up measurement | 3 months
  The change in psychological distress (CORE-OM) between the post-treatment measurement at the end of the 10-week intervention and the 3-month follow-up.
Change from baseline physiological and psychological symptoms (the Symptoms Check List-90; SCL-90) at 10-week post-treatment measurement | 10 weeks
  SCL-90 uses 90 items to measure nine primary symptomatic dimensions, including somatisation, obsessive-compulsiveness, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, and psychoticism. The level of distress is scored on a scale from 0 to 4. An average score of the 90 items is calculated, which represents the severity of the participant's symptoms, that is, the Global Severity Index (GSI).
Change from post-treatment physiological and psychological symptoms (the Symptoms Check List-90; SCL-90) at three-month follow-up measurement | 3 months
  The change in physiological and psychological symptoms (SCL-90) between the post-treatment measurement at the end of the 10-week intervention and the 3-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Raimo Lappalainen, Professor, Principal Investigator — University of Jyvaskyla

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hyvonen K, Pylvanainen P, Muotka J, Lappalainen R. The Effects of Dance Movement Therapy in the Treatment of Depression: A Multicenter, Randomized Controlled Trial in Finland. Front Psychol. 2020 Aug 12;11:1687. doi: 10.3389/fpsyg.2020.01687. eCollection 2020. PMID 32903394